CLINICAL TRIAL: NCT04535310
Title: Evaluation of Wear Experience With PRECISION1® Contact Lenses on Long Lens-wear Days
Brief Title: Wear Experience With Daily Contact Lenses Over a Long Day
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Alcon Research (Industry)
Responsible Party: Principal Investigator, Jennifer Fogt, Associate Professor Clinical, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0324
Record Dates: First submitted 2020-08-20; First posted 2020-09-01 (Actual); Results first posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Contact Lens
Keywords: Daily Disposable Contact Lens; Spherical Contact Lens; Soft Contact Lens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Daily Disposable Contact Lens (Experimental): All subjects are fit into Precision1® contact lenses. Subjects are requested to wear the lenses for a total of two weeks.
  Interventions: Device: Precision1® Daily Disposable Contact Lens

INTERVENTIONS:
Device: Precision1® Daily Disposable Contact Lens — Soft, spherical contact lens used to correct distance vision.

SUMMARY:
This study is evaluating the wear experience of a daily contact lens after 10, 12, 14, and 16 hours of lens wear.

ELIGIBILITY:
Inclusion Criteria:

* Must be a current spherical contact lens wearer with longs days of lens wear.
* Distance visual acuity of 20/25 or better with current contact lenses.
* Good general health (defined by medication use that has not changed within the last month and the absence of medical conditions or treatments that are deemed confounding to the data as determined by the PI).
* Recent eye exam within the past year.
* Must have a working smart phone and be willing to download an app and/or receive and respond to texts.
* Ability to give informed consent.
* Willing to spend time for the study. Subjects will be required to attend three study visits, wear contact lenses on days between study visits, and must respond to push-notifications and/or texts on a smart phone for 5 days between visits 2 and 3.

Exclusion Criteria:

* No current ocular inflammation or infection as assessed by the study investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fogt, OD, MS, Principal Investigator — The Ohio State University College of Optometry
Locations (1):
- The Ohio State University College of Optometry, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Daily Disposable Contact Lens
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daily Disposable Contact Lens
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.6 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Subjective Overall Comfort as Assessed Using the Visual Analog Scale (VAS)
Description: Subjective overall comfort as assessed using the Visual Analog Scale (VAS), with a scale of 0 to 100 with 0 being poor and 100 being excellent.
Time Frame: Up to 14 days
Population: participants
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Daily Disposable Contact Lens
Number analyzed (Participants) | 35
units on a scale | 93 [82.5 to 99]

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Daily Disposable Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-14): https://cdn.clinicaltrials.gov/large-docs/10/NCT04535310/Prot_SAP_001.pdf